CLINICAL TRIAL: NCT01460992
Title: Master Study for the MRI Compatibility of the EVIA/ENTOVIS Pacemaker in Combination With Safio S Pacemaker Lead
Brief Title: ProMRI AFFIRM Study of the EVIA/ENTOVIS Pacemaker With Safio S Pacemaker Leads
Acronym: ProMRIAFFIRM
Status: Completed | Type: Observational
Sponsor: Biotronik SE & Co. KG (Industry)
Responsible Party: Sponsor
Other Study IDs: 49
Record Dates: First submitted 2011-10-24; First posted 2011-10-27 (Estimated); Last update posted 2013-11-28 (Estimated); Status verified 2013-11

CONDITIONS: Cardiac Disease
Keywords: Pacemaker therapy; Magnetic Resonance Imaging (MRI); EVIA/ENTOVIS
MeSH Terms: conditions — Heart Diseases | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Pacemaker therapy: Patients with an EVIA/ ENTOVIS pacemaker device. See inclusion and exclusion criteria.
  Interventions: Procedure: Evia/Entovis pacemaker system under Magnetic Resonance Imaging (MRI) conditions

INTERVENTIONS:
Procedure: Evia/Entovis pacemaker system under Magnetic Resonance Imaging (MRI) conditions — patients will undergo an MRI scan for 30 minutes.
  Other Names: Evia/Entovis SR-T (single chamber with telemetry function), DR-T (dual chamber with telemetry function); Atrial/ventricular lead(s): Safio S 53 and S 60.; Safio S 45

SUMMARY:
This investigation is designed to demonstrate the clinical safety of the EVIA/ ENTOVIS pacemaker system when used under specific MRI conditions.

DETAILED DESCRIPTION:
In the past, MR scans were always contraindicated for pacemaker patients. If particular prerequisites and conditions are fulfilled, MR scans can now be conducted on patients with BIOTRONIK's EVIA/ENTOVIS pacemakers in combination with the Safio S pacemaker leads, scheduled to be part of this clinical study.

The specific MRI conditions for this investigation with the EVIA/ENTOVIS pacemaker family and Safio S pacemaker leads are defined in the study protocol

ELIGIBILITY:
Inclusion Criteria:

* Pacemaker system consisting solely of the EVIA/ENTOVIS pacemaker and Safio S pacemaker leads
* The pacemaker system has to be implanted, repositioned or exchanged at least 5 weeks prior to enrollment
* Age more than 18 years
* Understand the nature of the procedure
* Able and willing to complete MRI testing
* Able and willing to activate and use the Cardio Messenger
* Give written informed consent
* Able to complete all testing required by the clinical protocol
* Ability to measure atrial and/or ventricular pacing threshold(s)* (at 0.4 ms)
* All pacing thresholds do not exceed 2.0V @0.4ms.
* Available for follow-up visit at the investigational site
* Patient body height greater or equal to 140 cm
* Pectoral implantation
* The ascertained lead impedance is between 200 and 1500 Ohms.

Exclusion Criteria:

* No EVIA/ENTOVIS /Safio S pacemaker system implanted
* Pacing threshold(s) (at 0.4 ms) and sensing amplitudes are not measurable
* Meet one or more of the contraindications
* Being pregnant
* Have a life expectancy of less than three months
* Cardiac surgery already scheduled in the next three months
* Enrolled in another cardiac clinical investigation
* Have other medical implants that may interact with MRI, e.g. abandoned pacemaker/ICD leads, lead extensions, other active medical devices, non-MRI compatible devices (e.g. mechanical tricuspid valve)
* Have other metallic artifacts/components in body that may interact with MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients selected for participation should be from the investigator's general patient population according to the inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 121 (Actual)
Dates: Start 2012-03; Primary Completion 2013-10 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Primary hypothesis 1: MRI and pacing system related Serious Adverse Device Effect (SADE) free rate | 3 months
  MRI and pacing system related Serious Adverse Device Effect (SADE) Free-Rate is greater than 90%.
Primary hypotheses 2 and 3: pacing threshold rise (atrial and ventricular) | 1 month
  The atrial or ventricular MRI induced pacing threshold rise is not larger than or equal to 0.5 V between Pre-MRI and 1-month follow-up
Primary hypothesis 4: P-wave sensing attenuation | 1 month
  P-wave attenuation: P-wave amplitude decrease (between pre-MRI follow-up and 1-month follow-up) exceeding 50% or a P-wave amplitude at 1-month follow-up smaller or equal to 1.5 mV
Primary hypothesis 5: R-wave sensing attenuation | 1 month
  R-wave attenuation: R-wave amplitude decrease (between pre-MRI follow-up and 1-month follow-up) exceeding 50% or a R-wave amplitude at 1-month follow-up smaller or equal to 5.0 mV.

CONTACTS AND LOCATIONS:
Overall Officials: Aldo Rinaldi, Dr., Principal Investigator — Cardiology Department, St Thomas' Hospital Lambeth Palace Road London, SE1 7EH United Kingdom E-mail: Aldo.Rinaldi@gstt.nhs.uk
Locations (9):
- Allgemeines Krankenhaus Linz, Linz, Austria
- University Hospital Olomouc, Olomouc, Czechia
- Germany (5):
  - St. Gertrauden Krankenhaus, Berlin
  - Städtisches Klinikum Dresden-Friedrichstadt, Dresden
  - Uniklinik Leipzig, Leipzig
  - Diakoniekrankenhaus Mannheim, Mannheim
  - DRK Krankenhaus Neuwied, Neuwied
- Stadtspital Triemli, Zurich, Switzerland
- Cardiology Department, St Thomas' Hospital, London, United Kingdom

REFERENCES:
- [Derived] Bailey WM, Rosenthal L, Fananapazir L, Gleva M, Mazur A, Rinaldi CA, Kypta A, Merkely B, Woodard PK; ProMRI/ProMRI AFFIRM Study Investigators. Clinical safety of the ProMRI pacemaker system in patients subjected to head and lower lumbar 1.5-T magnetic resonance imaging scanning conditions. Heart Rhythm. 2015 Jun;12(6):1183-91. doi: 10.1016/j.hrthm.2015.02.010. Epub 2015 Feb 11. PMID 25680307